CLINICAL TRIAL: NCT04138810
Title: Assessment of Video-conference Technology for Post-operative Follow up in a Urogynecologic Population
Brief Title: Postoperative Virtual Clinical Encounters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Daniel Lee, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 830273
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post-op VCE (Experimental): As per standard of care, all subjects will be scheduled for a nursing clinical encounter 48-72 hours following discharge from the hospital from their surgery. The VCE group will conduct their encounter via the videoconference section of the MyChart mobile applications. At the end of this nursing encounter, the office nurse will schedule the patient for a 30 day postoperative visit within 4 to 6 weeks after their surgery.
  Interventions: Other: VCE; Other: Survey
- Office post-operative visits (Active Comparator): As per standard of care, all subjects will be scheduled for a nursing clinical encounter 48-72 hours following discharge from the hospital from their surgery. The traditional follow up group will receive a telephone call from the office nurse as is current standard of care. At the end of this nursing encounter, the office nurse will schedule the patient for a 30 day postoperative visit within 4 to 6 weeks after their surgery.
  Interventions: Other: Survey

INTERVENTIONS:
Other: VCE — Videoconference conducted according to a standard script which reviews the following key aspects of post-operative care: bowel functions, voiding functions, presence of vaginal bleeding, pain control, diet status, ambulatory status and any additional concerns. Standard post-operative instructions and precautions are reviewed as well.
  Arms: post-op VCE
Other: Survey — Measure of satisfaction regarding post-op visit.

SUMMARY:
Postoperative follow up is necessary following any surgical procedure and has been conducted in the same manner since the field of surgery began. The study will determine feasibility and patient satisfaction of innovative postoperative virtual clinical encounters utilizing mobile video conference technology for women undergoing pelvic reconstructive surgery through a randomized controlled trial.

DETAILED DESCRIPTION:
This will be a prospective randomized control study comparing postoperative virtual clinical encounters versus traditional in-office postoperative visits in women undergoing pelvic reconstructive surgery. The postoperative experiences of both groups will be assessed via surveys. Virtual Clinical Encounter Group: - Receive video-conference call from office nurse 48-72 hours post discharge from hospital - Receive video-conference call from fellow and/or attending physician approximately 30 days (4-6 weeks) from surgery -- Complete telephone survey one day later - Have in-office postoperative visit with fellow and/or attending physician approximately 90 days (10-12 weeks) from surgery -- Fill out surveys after office visit Traditional Office Group: - Receive telephone call from office nurse 48-72 hours post discharge from hospital - Have in-office postoperative visit with fellow and/or attending physician approximately 30 days (4-6 weeks) from surgery -- Complete telephone survey one day later - Have in-office postoperative visit with fellow and/or attending physician approximately 90 days (10-12 weeks) from surgery -- Fill out surveys after office visit

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery for pelvic organ prolapse
* Age greater than 18
* Access to a smartphone
* Access to high speed internet access (via 4G or 3G on their smartphone or high speed Wi-Fi)
* Signed up for MyPennMedicine web portal
* Ability to download MyChart mobile application
* Pennsylvania Hospital Subject: NJ or PA resident, HUP & Presbyterian Hospital Subject: PA resident

Exclusion Criteria:

* Pregnancy
* Inability to read, speak or understand English
* Isolated midurethral sling procedure
* Extraperitoneal vaginal colpopexy with Uphold mesh

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee DD, Arya LA, Andy UU, Harvie HS. Video Virtual Clinical Encounters Versus Office Visits for Postoperative Care After Pelvic Organ Prolapse Surgery: A Randomized Clinical Trial. Female Pelvic Med Reconstr Surg. 2021 Jul 1;27(7):432-438. doi: 10.1097/SPV.0000000000000909. PMID 32604202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post-op VCE | Office Post-operative Visits
Started | 27 | 27
Completed | 26 | 26
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Subject cancelled surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-op VCE | Office Post-operative Visits | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (10.9) | 58.0 (11.3) | 58.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 23 | 44
  Black | 3 | 3 | 6
  Hispanic | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction Via the Patient Satisfaction Questionnaire -18
Description: PSQ-18 is a validated eighteen item patient satisfaction questionnaire that has been utilized across diverse healthcare settings. It measures satisfaction across the following domains: general satisfaction, technical quality of care, interpersonal manner of healthcare provider, communication, financial aspects of care, time spent with healthcare provider and accessibility/convenience of care. Total scores range from 18 to 90, with higher scores indicating higher patient satisfaction.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-op VCE | Office Post-operative Visits
Number analyzed (Participants) | 26 | 26
score on a scale | 80.7 (2.6) | 81.2 (2.8)
Statistical Analysis 1: Comparison: Post-op VCE vs Office Post-operative Visits; Test type: Non-Inferiority — We defined the non-inferiority margin to be 5 points which with a sample of size of 25 women per arm would mean we would have a type I error rate of 0.05 and a power of 0.80; Mean Difference (Net) = 0.46, 95% CI 2-sided [-1.95 to 1.03]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject for 90 days, from date of surgery to 90 days post-surgery.
Description: For this protocol, only adverse events that were related to the participant's participation in research were collected.
Arm/Group | Post-op VCE | Office Post-operative Visits
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04138810/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04138810/ICF_001.pdf